CLINICAL TRIAL: NCT06797050
Title: A Story for Pepper and Nao: Applying the Learning by Teaching Paradigm in Children With Patterns of Neuromotor Impairment
Brief Title: A Story for Pepper & Nao
Acronym: LbyT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: IRCCS Eugenio Medea (Other); Fondazione Mondino (Other); University of Florence (Other)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, Professor, IRCCS Fondazione Stella Maris
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LbyT
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Children and Adolescents With Neuromotor Impairment
Keywords: Learning by teaching; Social robot; Children; Neuromotor impairment; Executive Functions; Engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental Group) (Experimental): The experimental group, following an initial assessment, will carry out the training. The child will be asked to help the social robot, which will provide relational and learning feedback, to reorder sequences of images from figurative stories, in order to create a story that respects temporal or causal links, or motor actions of increasing complexity, according to the Learning by Teaching paradigm. The images, which will appear on the social robot's tablet, will be presented with increasing complexity and numerosity, and in the case of difficulty, facilitation will be provided in such a way as to encourage 'mistake-free' learning. In each session (approx. 20-25), on a bi-weekly basis, will be an operator will be present. The engagement experienced by the child on an emotional, behavioural and cognitive level will be measured. A second assessment is scheduled at the end of the training and a third after about 4 months.
  Interventions: Device: Training in reordering figurative stories with a social robot through the Learning by Teaching approach
- Group 2 (Control group) (No Intervention): After an initial assessment, children assigned to the control group will be asked to continue with what they normally do (standard care). Only after a period of about four months, following the second assessment they will begin treatment with the social robot, described for the experimental group.

INTERVENTIONS:
Device: Training in reordering figurative stories with a social robot through the Learning by Teaching approach — A test session of the 'picture sequencing' task with the social robot is planned. The selected children will undergo an initial neuropsychological, motor and school learning assessment and will be divided into Group 1 and Group 2: Group 1 (Experimental) will be offered training with the social robot, while Group 2 (Control) will continue standard care. Both groups will be re-evaluated after approximately about 4 months. After which Group 2 will be able to start treatment. After about 4 months, the children in both groups will again undergo the planned assessments. During the training, the child will be asked to help the social robot to reorder sequences of pictures from figurative stories in order to create a story that respects temporal or causal links, or motor actions of increasing complexity, according to the Learning by Teaching paradigm.
  Arms: Group 1 (Experimental Group)

SUMMARY:
The aim of the present study is to improve cognitive processes that are frequently impaired in children characterised by neuromotor impairment, such as the skills of visual-perceptual analysis and selective attention, working memory, narrative organisation, logical-inferential reasoning and motor planning. For this purpose, a task of reordering figurative stories and action sequences, which include the aforementioned processes, will be used through an innovative Learning by Teaching training paradigm with a social robot. Furthermore, the study aims to verify the children's level of behavioural, cognitive and emotional engagement during the interaction with the social robot and to test the generalisation effects of the intervention on other processes, such as working memory, inhibition and planning.

DETAILED DESCRIPTION:
The use of social robots in children with Neurodevelopmental Disorders and Disabilities is becoming increasingly common in both educational and clinical settings. Several studies have shown that the presence of social robots during learning can increase children's engagement, consequently improving academic achievement, as the presence of the robot appears to positively influence attention, satisfaction, and engagement in the proposed activities. Engagement is a complex component that includes emotional, cognitive, and behavioral aspects. The emotional component concerns the emotions felt during the activity, the cognitive component involves attention and active participation, and the behavioral component refers to the user's proactivity and adaptability in the interaction. An innovative approach of using social robots is the Learning by Teaching paradigm, where children teach the robots, thus promoting their sense of self-efficacy and motivation, as well as the ability to put themselves in each other's shoes (Theory of Mind). This method helps develop Executive Functions, such as planning, problem solving and reasoning, which are crucial to various aspects of daily life. Skills that are often vulnerable in children with Neurodevelopmental Disorders and Disabilities, consequently associating with poor performance in school learning, including text comprehension and production, which require good decoding skills, logical reasoning, selective attention, interference control, working memory and metacognitive strategies. Several studies have also shown that children with neuromotor impairment pictures, such as Motor Coordination Disorder (DCD) or Cerebral Palsy (CP), often have difficulties in motor planning skills, which become worse with the specificity of the motor problem. A "picture sequencing" task, which involves arranging pictures in order to create a finalized story or movement, can support multiple higher cognitive processes, such as working memory, attention, reasoning, and planning. This task, embedded in the Learning by Teaching paradigm with a social robot, could amplify the development of these processes due to the high levels of engagement and the requirement to take on the robot's role as teacher. In order to test the effectiveness of the treatment in improving the skills of visual-perceptual analysis, selective attention, working memory, narrative organization, logical-inferential reasoning and motor planning, 80 children with neuromotor difficulties will be randomly assigned to either the Experimental Group, which will immediately begin treatment with the social robot for about 4 months on a biweekly schedule, or to the Control Group, which will begin training after about 4 months. In addition, the study aims to test the children's level of behavioral, cognitive and emotional engagement during interaction with the social robot, through the use of sensors, eye-tracking and video cameras; as well as to test the generalization effects of the intervention on other processes, such as working memory, inhibition and planning.

ELIGIBILITY:
Inclusion Criteria:

* Children characterized by neuromotor impairment
* Presence of at least one cognitive index >70 at WISC-IV or WISC V
* Age between 7 and 16 years at the time of recruitment

Exclusion Criteria:

* Severe neurological, motor, or sensory deficit such as to preclude the feasibility of training
* Psychiatric comorbidity such as to preclude the feasibility of training

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
score of Picture Arrangement subtest at WISC-III | 1-16 months
  In this study, examiners will administer the Picture Arrangement subtest of the WISC-III (Wechsler, 1991), in which children are presented with a series of cards in random order that need to be placed in the correct order to tell a meaningful story.
score of a Motor Planning test | 1-16 months
  In this study, examiners will assess changes in motor planning skills as measured by a purpose-built test.

SECONDARY OUTCOMES:
score of Corsi block-tapping subtest at the BVS-Corsi | 1-16 months
  In this study, examiners will administer the Corsi block-tapping subtets at the BVS-Corsi (Mammarella et al., 2008), to evaluate visuo-spatial short term and working memory. The child is asked to retrieve a sequences previously seen by the examiner by tapping blocks with the preferred finger following the same order for the forward condition or reversing the order for the backward condition.
score of Tower of London test | 1-16 months
  In this study, examiners will administer the Tower of London test (Fancello et al., 2006; Gugliotta et al., 2009) to assesses the planning ability. There are three pegs of different lengths, into which three marbles are threaded the subject has to move these marbles in a certain number of moves in order to achieve the configuration indicated by the examiner
score of the Sustained Attention subtest at the Leiter-3 | 1-16 months
  In this study, the examininers will use the Sustained Attention subtest at the Leiter International Performance Scale Leiter-3 (Roid et al., 2013), which assesses visual attention and consist of repetitive barrage tasks to be performed in a predefinited time.
score of Behaviour Rating Inventory of Executive Function for parents (BRIEF-2) | 1-16 months
  In this study, examiners will administer the BRIEF-2 questionnaire (Gioia et al., 2015). This questionnaire is filled by the parents/legal guardians and dives into everyday bahaviour associated with specific domains of the Exefutive Functions (i.e., mental processes that enable us to plan, focus attention, remember instructions). Parents rate items on a three-point scale ranging from 1 (never) to 3 (often)
score of Inhibition subtest at the NEPSY-II | 1-16 months
  In this study, the examiners will assess the Inibition subtest at the NEPSY-II (Urgesi et al., 2011), in which the child will be asked to naimed different shapes according to examiners instructions.
score of Verbal Fluency subtest at the NEPSY-II | 1-16 months
  In this study, the examiners will assess the Verbal Fluency subtest at the NEPSY-II (Urgesi et al., 2011), which evaluates cognitive flexibility in a word production task within a specific semantic or phonemic category.
score of Animal Sorting subtest at the NEPSY-II | 1-16 months
  In this study, examiners will assess the Animal Sorting subtest at the NEPSY-II (Urgesi at al., 2011). This subtest is designed to assess the ability to formulate basic concepts, to transfer those concepts into action (sort into categories), and to shift set from one concept to another. The child sorts cards into two groups of four cards each using various self-initiated sorting criteria.
score of Go/No-Go subtest at the TeleFE | 1-16 months
  In this study, the examiners will assess Go/No-Go subtest at the TeleFE (Cooperativa Sociale Anastasis), that is a web platform for the multidimensional assessment of Executive Functions. In the Go/No-Go subtest children are asked to press a button when the target stimulus.
score of Text comprehension test at Prove MT-3, MT Avanzate and MT 16-19 | 1-16 months
  In this study, the examiners will assess the text comprehension ability trhough Prove MT-3, MT Avanzate and MT 16-19(Cornoldi et al., 2016 and 2022). In this test, the child is asked to read a text and answer some questions related to it in order to assess text comprehension.
score of Invent a story task | 1-16 months
  In this study, the examiners will assess the Invent a story task, in which children are required to orally tell a invented story in order to assess narrative production
score of TVPS-4 test | 1-16 months
  In this study, the examiners will assess Test of Visual Perceptual Skills-4th Edition (TVPS-4) (Martin A., 2017) to evaluate visual-perceptual strenghts and weaknesses.
score of DCDDaily-Q | 1-16 months
  In this study, examiners will administer the DCDDaily-Q (Van Der Linde et al., 2014). The DCDDaily-Q is a parental questionnaire to address children's performance in Activities of Daily Living (ADL).
score of Abilhand/Abilhand kids questionnaire | 1-16 months
  In this study, the examiners will administer the Abilhand/Abilhand kids questionnaire (Penta et al., 2001; Arnould et al., 2004), that is an interview-based assessment of a patient-reported measure of the perceived difficulty in using their hand to perform manual activities in daily activities.
Evaluation of engagement levels during interaction with the social robot | 1-16 months
  During the child's interaction with the social robot, three different levels of engagement will be measured: emotional through wearable sensors (e.g. Fitbit, Shimmer or similar); cognitive through eye-gazing extracted from video recordings using software such as DeepGaze or Gaze360 to assess attentional maintenance; and behavioural through video analysis of the child's postures, amount of movements, and verbal expressions. Questionnaires are also planned to assess the degree of acceptability and feasibility of the activity with the social robot

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Eugenio Medea, Bosisio Parini, Lecco
  - IRCCS Istituto Neurologico Naz.le C.Mondino, Pavia, Pavia
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wotherspoon J, Whittingham K, Sheffield J, Boyd RN. Cognition and learning difficulties in a representative sample of school-aged children with cerebral palsy. Res Dev Disabil. 2023 Jul;138:104504. doi: 10.1016/j.ridd.2023.104504. Epub 2023 Apr 24. PMID 37099882
- [Background] Fuglerud KS, Solheim I. The Use of Social Robots for Supporting Language Training of Children. Stud Health Technol Inform. 2018;256:401-408. PMID 30371501
- [Background] Fluss J, Lidzba K. Cognitive and academic profiles in children with cerebral palsy: A narrative review. Ann Phys Rehabil Med. 2020 Oct;63(5):447-456. doi: 10.1016/j.rehab.2020.01.005. Epub 2020 Feb 19. PMID 32087307
- [Background] Fiorini L, D'Onofrio G, Sorrentino A, Cornacchia Loizzo FG, Russo S, Ciccone F, Giuliani F, Sancarlo D, Cavallo F. The Role of Coherent Robot Behavior and Embodiment in Emotion Perception and Recognition During Human-Robot Interaction: Experimental Study. JMIR Hum Factors. 2024 Jan 26;11:e45494. doi: 10.2196/45494. PMID 38277201
- [Background] Fiorini L, De Mul M, Fabbricotti I, Limosani R, Vitanza A, D'Onofrio G, Tsui M, Sancarlo D, Giuliani F, Greco A, Guiot D, Senges E, Cavallo F. Assistive robots to improve the independent living of older persons: results from a needs study. Disabil Rehabil Assist Technol. 2021 Jan;16(1):92-102. doi: 10.1080/17483107.2019.1642392. Epub 2019 Jul 22. PMID 31329000
- [Background] Dionne E, Bolduc ME, Majnemer A, Beauchamp MH, Brossard-Racine M. Academic Challenges in Developmental Coordination Disorder: A Systematic Review and Meta-Analysis. Phys Occup Ther Pediatr. 2023;43(1):34-57. doi: 10.1080/01942638.2022.2073801. Epub 2022 May 24. PMID 35611495
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Di Lieto MC, Pecini C, Castro E, Inguaggiato E, Cecchi F, Dario P, Cioni G, Sgandurra G. Empowering Executive Functions in 5- and 6-Year-Old Typically Developing Children Through Educational Robotics: An RCT Study. Front Psychol. 2020 Feb 5;10:3084. doi: 10.3389/fpsyg.2019.03084. eCollection 2019. PMID 32116879
- [Background] https://doi.org/10.1007/s11145-021-10205-x
- [Background] Belpaeme T, Kennedy J, Ramachandran A, Scassellati B, Tanaka F. Social robots for education: A review. Sci Robot. 2018 Aug 15;3(21):eaat5954. doi: 10.1126/scirobotics.aat5954. Epub 2018 Aug 15. PMID 33141719
- [Background] Beani E, Filogna S, Martini G, Barzacchi V, Ferrari A, Guidi E, Menici V, Cioni G, Sgandurra G. Application of Virtual Reality Rehabilitation System for the assessment of postural control while standing in typical children and peers with neurodevelopmental disorders. Gait Posture. 2022 Feb;92:364-370. doi: 10.1016/j.gaitpost.2021.12.008. Epub 2021 Dec 10. PMID 34923256
- [Background] Adams IL, Lust JM, Wilson PH, Steenbergen B. Compromised motor control in children with DCD: a deficit in the internal model?-A systematic review. Neurosci Biobehav Rev. 2014 Nov;47:225-44. doi: 10.1016/j.neubiorev.2014.08.011. Epub 2014 Sep 1. PMID 25193246